CLINICAL TRIAL: NCT07067034
Title: The Riddikulus Nursing Intervention: A Brief, Nurse-Led Intervention to Reduce Student Anxiety in a Randomized Controlled Study
Brief Title: Nurse-Led Intervention (Riddikulus) to Reduce Anxiety in University Students
Acronym: RNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege Miray Topcu (Other)
Responsible Party: Sponsor-Investigator, Ege Miray Topcu, Research Assistant Ege University, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-2T/44; 1919B012205498 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Nurse-led Supportive Care; Nursing Interventions
Keywords: Anxiety; University Students; Psychosocial Nursing Intervention; brief intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received the Riddikulus Nursing Intervention, or the control group, which received no intervention. Each participant remained in their assigned group throughout the study. Anxiety levels were assessed at three time points: before, immediately after, and at follow-up.
Who Masked: Care Provider
Masking Description: Group allocation was blinded to the investigators and care providers during participant assignment. Randomization codes were prepared by an independent person who did not take part in data collection or intervention delivery. After group assignment, participants and researchers were aware of the allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riddikulus Intervention Group (Experimental): Participants in this group received a one-session, metaphor-based psychosocial nursing intervention. The intervention involved identifying anxiety-related personal metaphors and restructuring them into less distressing or humorous mental images under the guidance of a trained academic nurse.
  Interventions: Behavioral: Ridikullus Nursing İntervention
- control group (No Intervention): Participants in this group received no intervention. They completed the same outcome measures at the same time points as the intervention group, but did not receive any psychological or nursing-based session.

INTERVENTIONS:
Behavioral: Ridikullus Nursing İntervention — A one-session, nurse-led psychosocial intervention designed to reduce anxiety in university students. Participants identified personal metaphors related to their anxiety and were guided to reconstruct them into less distressing, humorous, or calming mental images. The intervention was delivered in a structured format by an academic nurse trained in therapeutic communication
  Arms: Riddikulus Intervention Group

SUMMARY:
This randomized controlled trial investigates the effectiveness of the Riddikulus Nursing Intervention, a brief, low-cost, nurse-led strategy designed to reduce anxiety levels in university students. The intervention uses metaphor-based reflection and creative emotional flexibility techniques in a single-session format. A total of 36 participants were randomly assigned to intervention and control groups. Anxiety levels were measured using the Visual Analog Scale (VAS) and the Beck Anxiety Inventory (BAI) before and after the intervention. The study aims to evaluate whether this innovative, easily applicable approach can significantly reduce short-term perceived anxiety in young adults.

DETAILED DESCRIPTION:
This study investigates the effectiveness of a novel, low-cost, nurse-led psychological intervention called the Riddikulus Nursing Intervention, designed to reduce anxiety levels in university students with moderate anxiety. The intervention was inspired by a metaphorical coping scene from the Harry Potter film series and structured as a single-session, creative, and non-pharmacological approach. During the intervention, participants were asked to generate personal metaphors related to their anxiety and were guided in restructuring these metaphors into less distressing, humorous, or soothing mental images. The process was facilitated by an academic mentor trained in therapeutic communication.

The study was conducted at the School of Foreign Languages of Ege University between December 2023 and June 2024. A total of 1100 students were invited, and 549 agreed to participate. Among students with moderate levels of anxiety, 36 participants were included and the study was completed with them. These participants were randomly assigned to intervention (n=17) and control (n=19) groups. Anxiety levels were assessed at three time points-pre-intervention, post-intervention, and follow-up-using the Visual Analog Scale (VAS) and the Beck Anxiety Inventory (BAI). Data analysis was performed with SPSS 25.0, and participant flow was reported using the CONSORT diagram.

The results revealed a statistically significant reduction in VAS anxiety scores within the intervention group, with a large effect size. However, no significant differences were observed in BAI scores between the groups over time. These findings suggest that the Riddikulus Intervention may be particularly effective in reducing short-term, perceived anxiety in young adults. Participants also reported subjective improvements in emotional state and metaphor transformation following the session.

This study highlights the feasibility and promise of brief, creative, nurse-led interventions for managing moderate anxiety in university settings. Further research with larger sample sizes, repeated sessions, digital delivery formats, and long-term follow-up assessments is recommended to validate and expand upon these findings.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student at the School of Foreign Languages, Ege University during the study period
* No history of repeating an academic year
* No hearing or visual impairments
* No prior psychiatric diagnosis
* Not currently undergoing psychiatric treatment or therapy
* A score between 16 and 25 on the Beck Anxiety Inventory (BAI), indicating moderate anxiety
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Failure to attend the intervention session
* Withdrawal of voluntary consent at any time

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level measured by Beck Anxiety Inventory (BAI) | Baseline, Immediately Post-Intervention, 4-Week Follow-Up
  The Beck Anxiety Inventory (BAI) was used to assess clinical anxiety symptoms. It is a 21-item self-report instrument, with higher total scores reflecting higher levels of anxiety. The Beck Anxiety Inventory (BAI) ranges from 0 to 63, with higher scores indicating greater levels of anxiety
Change in anxiety level measured by Visual Analog Scale (VAS) | Baseline, Immediately Post-Intervention
  Anxiety was assessed using a 0-10 Visual Analog Scale (VAS), with higher scores indicating greater anxiety. Measurements were taken before the intervention, immediately after, and two weeks following the session. Lower scores reflect reduced levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including age, gender, Beck Anxiety Inventory (BAI) scores, and Visual Analog Scale (VAS) scores collected at baseline, immediately post-intervention, and 4-week follow-up will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of primary results
Access Criteria: Qualified researchers who provide a methodologically sound proposal may request access to de-identified individual participant data, the study protocol, and the statistical analysis plan. Data will be shared via secure institutional email after obtaining approval from the principal investigator and the ethics committee.